CLINICAL TRIAL: NCT06287983
Title: Effect of Inspiratory Muscle Training on Respiratory Functions and Exercise Capacity in Patients With Ankylosing Spondylitis Receiving Anti-TNF Therapy: Randomized Controlled Study.
Brief Title: Effect of Inspiratory Muscle Training on Respiratory Functions and Exercise Capacity
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kayseri City Hospital (Other Government)
Responsible Party: Principal Investigator, Havva Talay Çalış, professor doctor, Kayseri City Hospital
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: KayseriCHIMT001
Record Dates: First submitted 2024-02-24; First posted 2024-03-01 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Ankylosing Spondylitis
MeSH Terms: conditions — Spondylitis, Ankylosing

STUDY DESIGN:
Intervention Model Description: A total of 44 patients were randomly divided into 2 groups using the sealed envelope randomization method. The exercise program will be applied to both groups 3 sessions a week for 60 minutes for 6 weeks. Inspiratory muscle training will also be added to the intervention group. Patients included in the study; At weeks 0, 6, 12 and 24, BASDAI (Bath Ankylosing Spondylitis Disease Activity Index), BASFI (Bath Ankylosing Spondylitis Functional Index), ASQoL (The Ankylosing Spondylitis Quality of Life), Modified Borg Scale, Visual Analog scale (VAS) and maximum Dyspnea measurement during exercise, 6-minute walk test, chest expansion measurement and respiratory function test (spirometry) will be evaluated.
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EXERCISE GROUP (Experimental): The Sample Spondylitis Exercise Program
  Interventions: Other: The Sample Spondylitis Exercise Program
- EXERCISE+ Inspiratory muscle trainer (IMT) GROUP (Active Comparator): The Sample Spondylitis Exercise Program Inspiratory muscle training will also be added to the intervention group.
  Interventions: Device: Inspiratory Muscle Trainer (IMT) (POWERbreathe Medic Classic); Other: The Sample Spondylitis Exercise Program

INTERVENTIONS:
Device: Inspiratory Muscle Trainer (IMT) (POWERbreathe Medic Classic) — Inspiratory muscle training will be started at an intensity of 50% of the patient's measured PIMAX value and will be increased by 2 cm/H20 per day according to patient tolerance, and will be applied for a total of 6 weeks / 5 days per week / 3 sessions per day / 10 breaths per session.
  Arms: EXERCISE+ Inspiratory muscle trainer (IMT) GROUP
Other: The Sample Spondylitis Exercise Program — The Sample Spondylitis Exercise Program recommended by the Spondylitis Association of America will be translated into Turkish and each exercise will be applied in 3*10 sets. The exercise program will be applied to both groups, 3 sessions a week for 60 minutes for 6 weeks.

SUMMARY:
In this study, we aimed to evaluate the effect of Anti- tumor necrosis factor (TNF) treatment on pulmonary functions in patients with AS and to evaluate the pulmonary functions and exercise performance of patients by adding inspiratory muscle training to spinal mobility exercises in patients with AS using Anti-TNF. We also aimed to investigate the relationship between these parameters and disease activity, spinal mobility and quality of life.

DETAILED DESCRIPTION:
Patients diagnosed with AS who applied to outpatient clinic, received anti- tumor necrosis factor (TNF) treatment for at least 6 months and have been evaluated will be included in the study.

Patients who agree to participate in the study will be asked to sign a consent form. At the beginning, all patients' name-surname, age, height, body weight, body mass index, smoking-alcohol use, profession, marital status, education, duration of ankylosing spondylitis disease, history of corticosteroid use, presence of systemic and extra-articular involvement, medications used and additional diseases will be questioned and recorded in their files.

It was planned to include 30 male and 14 female patients in the study by calculating the female/male ratio of patients diagnosed with As who applied to hospital in the last year and in line with the literature. A total of 44 patients will be randomly randomized into 2 groups using the sealed envelope randomization method. The exercise program will be applied to both groups, 3 sessions a week for 60 minutes for 6 weeks.

The Sample Spondylitis Exercise Program recommended by the Spondylitis Association of America will be translated into Turkish and each exercise will be applied in 3*10 sets.

Inspiratory muscle training will also be added to the intervention group.

Inspiratory muscle training will be started at an intensity of 50% of the patient's measured PIMAX value and will be increased by 2 cm/H20 per day according to patient tolerance, and will be applied for a total of 6 weeks / 5 days per week / 3 sessions per day / 10 breaths per session.

Patients included in the study were evaluated with BASDAI (Bath Ankylosing Spondylitis Disease Activity Index), BASFI(Bath Ankylosing Spondylitis Functional Index), ASQoL(The Ankylosing Spondylitis Quality of Life), Modified Borg Scale, measurement of dyspnea at maximum exercise with Visual Analog Scale (VAS), 6-minute walk test, chest expansion measurement and respiratory function test (spirometry) at 0, 6, 12 and 24 weeks will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with ankylosing spondylitis according to the Modified New York Criteria
* Patients with BASDAI score <4.1 who received Anti-TNF therapy for at least 6 months
* Patients whose maximum inspiratory pressure value is <80% in the Pulmonary Function Test
* Patients who had a cardiac examination within the last year and no cardiac pathology was detected.

Exclusion Criteria:

* The patient has a serious mental disorder
* Presence of neurological and pulmonary disease that would prevent the patient from using the PFT device
* Presence of uncontrolled hypertension
* Presence of uncontrolled diabetes
* Presence of uncontrolled cardiac arrhythmia
* Uncontrolled heart failure
* High-risk unstable angina and all acute cardiac diseases (acute myocardial infarction, acute endocarditis, myocarditis or pericarditis)
* Symptomatic severe aortic stenosis
* Acute pulmonary embolism or pulmonary infarction
* Severe pulmonary hypertension
* Presence of systemic infection or malignancy
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-05-15 (Estimated)

PRIMARY OUTCOMES:
Respiratory function test (Spirometry) | before treatment (day 0), after treatment (week 6), after treatment (week 12), after treatment (week 24)
  Spirometry is the most commonly used respiratory function test (PFT). It is a physiological test based on measuring the flow or volume changes that occur during breathing as a derivative of time. The standard maneuver used during spirometry is also called the forced expiratory maneuver; It consists of rapid and deep inspiration followed by maximal expiration at the level of total lung volume. The spirometry test to be evaluated must comply with the previously defined spirometry test performance standards, acceptability and repeatability criteria. In the study, the most frequently measured spirometric parameters with forced expiration maneuver were; vital capacity (VC), forced vital capacity (FVC), forced expiratory volume (FEV), maximum inspiratory pressure (PImax) and maximum expiratory pressure (Pemax) to evaluate respiratory muscle strength will be checked.

SECONDARY OUTCOMES:
Bath Ankylosing Spondylitis Disease Activity Index (BASDAI): | before treatment (day 0), after treatment (week 6), after treatment (week 12), after treatment (week 24)
  It evaluates disease-specific symptoms such as fatigue, spinal and peripheral joint pain, swelling and morning stiffness and is interpreted on a score ranging from 0-10. An increase in the score indicates an increase in disease activity. It is a reliable and sensitive index developed to evaluate disease activity and progression.
Bath Ankylosing Spondylitis Functional Index (BASFI) | before treatment (day 0), after treatment (week 6), after treatment (week 12), after treatment (week 24)
  It is a fast and easy-to-apply, sensitive and reliable index developed to determine and monitor the functional status of patients with AS. It consists of 10 questions that evaluate patients' abilities to bend, reach, stand, change positions, climb stairs, and cope with activities of daily living. For each question, the final score is obtained by dividing the total score by 10 using VAS in the range of 0-10 cm.
Ankylosing Spondylitis Quality of Life Questionnaire (ASQoL) | before treatment (day 0), after treatment (week 6), after treatment (week 12), after treatment (week 24)
  ASQoL is the most widely used, valid and reliable questionnaire to evaluate the quality of life in AS. In this survey, which consists of eighteen questions, patients are asked to answer yes or no to each question. '0' points are taken for a no answer and '1' point is taken for a yes answer. Total score varies between 0-18. High scores indicate serious impairments in quality of life.
Modified Borg Scale | before treatment (day 0), after treatment (week 6), after treatment (week 12), after treatment (week 24)
  It is a scale frequently used to evaluate the severity of exertion dyspnea and resting dyspnea severity. It consists of ten items that describe the severity of dyspnea according to its degree. Defining the severity of dyspnea in the Modified Borg Scale makes it easier for patients to apply.
Measurement of dyspnea at maximum exercise with the Visual Analog Scale (VAS) | before treatment (day 0), after treatment (week 6), after treatment (week 12), after treatment (week 24)
  Visual Analog Scale (VAS) is a scale applied by marking with a pencil on a horizontal or vertical line of one hundred millimeters. There is no dyspnea at the 0 mm point of this line, and the most severe dyspnea is at the 100 mm point. The patient marks the severity of the current respiratory distress on the scale using these two degrees as criteria. Scoring is done by measuring the marked point with the help of a tape measure. Most of the studies conducted to date indicate that VAS is a reliable scale that can be used to evaluate the severity of dyspnea, and that it is even sensitive to minute changes in the severity of dyspnea.
6-minute walk test (6MWT) | before treatment (day 0), after treatment (week 6), after treatment (week 12), after treatment (week 24)
  It is a frequently used test in cardiopulmonary rehabilitation to monitor exercise capacity and treatment effectiveness. The patient should rest by sitting in a chair for 15 minutes before the test and wear appropriate shoes and comfortable clothing. Calculate the distance walked by the patient at their own walking pace in 6 minutes, preferably in a 30-meter long corridor. If the patient's O2 saturation (sO2) is <88%, the test should be performed with O2 support.
Chest expansion measurement | before treatment (day 0), after treatment (week 6), after treatment (week 12), after treatment (week 24)
  Chest expansion is measured at the fourth intercostal space. The patient is asked to exhale all the air in his lungs and then take deep inspiration. As a result of deep inspiration, the expansion around the chest is recorded in centimeters.

CONTACTS AND LOCATIONS:
Overall Officials: Serap Tomruk Sütbeyaz, Prof, Study Director — Saglik Bilimleri Universitesi; Esra Yaprak tas, Principal Investigator — Saglik Bilimleri Universitesi
Locations (1):
- Health Sciences University, Kayseri Medicine Faculty, Kayseri City Hospital, Kayseri, Turkey (Türkiye)